CLINICAL TRIAL: NCT07302308
Title: Action Outcome Latencies as a Measure of Sense of Agency in Functional Movement Disorders.
Status: Not yet recruiting | Type: Observational
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Aditya Murgai, Assistant Professor, Western University, Canada
Other Study IDs: Action outcome latencies
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Functional Movement Disorder
Keywords: functional movement disorder; sense of agency; judgment of agency
MeSH Terms: conditions — Conversion Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Functional Movement Disorder
- Controls: Healthy subjects

SUMMARY:
Functional movement disorders (FMD) are among the most common neurological conditions seen in clinical practice, yet they are poorly understood and often misdiagnosed. Impaired self-agency, the sense of controlling one's actions, is a key feature of FMD. Studies using functional MRI have shown reduced activation and connectivity in the right inferior parietal lobule, a region associated with agency.

The sense of agency consists of two components: the feeling of agency, which is an implicit, low-level sense of control over voluntary actions, and the judgment of agency, which is the conscious attribution of actions to oneself. While the feeling of agency is often measured using intentional binding tasks, judgment of agency is assessed using self-reported scales. While studies have explored intentional binding as a measure of implicit agency in FMD, few have systematically investigated judgment of agency. This study aims to fill this gap by introducing a novel approach that quantitatively evaluates judgment of agency in FMD patients using action-outcome latencies as an objective metric.

DETAILED DESCRIPTION:
Objective: The objective of this study is to investigate the differences between patients with FMD and healthy controls in perceiving visual and auditory outcomes as consequences of their actions. This will be assessed by measuring their judgment of agency through action-outcome latencies.

ELIGIBILITY:
Inclusion criteria for patients: Inclusion criteria for patients:

1. Diagnosed with clinically definite functional movement disorder
2. Age >18 years.
3. Able to read and understand English.

Inclusion criteria for healthy subjects:

1. Age >18 years.
2. Able to read and understand English

Exclusion criteria for patients:

1. Moderate to severe action tremor in the dominant hand limiting the ability to perform the task.
2. Upper limb peripheral neuropathy.
3. Unable to read and understand English.

Exclusion criteria for healthy subjects:

1. Unable to read and understand English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: movement disorder clinic
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
SA Index | Day 1
  Latencies values corresponding to positive ("YES") responses will be extracted. SA (Sense of Agency) Index will be computed by multiplying the 90th percentile latencies by the number of positive responses below this latency threshold and then dividing the result by the total number of responses (positive, negative and unsure) occurring below the same threshold.
Latencies | Day 1
  The 90th percentile of latency values among trials with positive ("YES") responses.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
At this time, IPD will not be shared due to confidentiality concerns.